CLINICAL TRIAL: NCT02381574
Title: French Lumbar Total Disk Replacement Observational Study (FLTDR Observational Study)
Brief Title: French Lumbar Total Disk Replacement Observational Study
Acronym: PTDL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medtronic France SAS (Industry)
Collaborators: DePuy Synthes (Industry); LDR Médical (Unknown)
Responsible Party: Sponsor
Other Study IDs: PTDL
Record Dates: First submitted 2015-02-18; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Lumbar Total Disk Replacement
Keywords: Lumbar Total Disk Replacement

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objective:

To evaluate the rate of re-operation during the first 5 years following the fitting of lumbar total disk replacement at the operated level and / or floors above and / or underlying, whatever the reasons

DETAILED DESCRIPTION:
Secondary objectives:

The secondary objectives are:

* Describe the reasons for re-interventions operated floor and / or (x) level (s) adjacent (s)
* Describe the evolution of the function with the functional Oswestry score
* Describe the evolution of lumbar radicular pain by visual analog scale (VAS)
* Describe the evolution of the quality of life assessed by the SF12 score
* Describe the evolution of work status
* Describe patient satisfaction
* Describe the complications (intraoperative, early postoperative (within 3 months of surgery), late, death)

ELIGIBILITY:
Inclusion Criteria:

* Patient who needs, according to his surgeon, a PTDL placement and has given his consent for the PTDL placement
* Patient who agrees to participate in the observational study after information by the surgeon
* Patient living in France and having the ability to respond alone to the questionnaire

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Analysis of the first 600 patients implanted with a PTDL (first 200 prostheses implanted for each laboratory involved in the observational study): Medtronic, LDR Médical et Synthes SAS) during an estimated inclusion period from 6 to 18 months and a follow-up period of 5 years.
  An additional follow-up from 3 to 5 years will be envisaged in a protocol amendment if requested by Authorities.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-06; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of re-intervention during the first 5 years after fitting of total disk replacement | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard SCHROEDER, Study Chair — SNITEM
Locations (69):
- France (69):
  - Clinique Herbert, Aix-les-Bains
  - Clinique HERBERT, Aix-les-Bains
  - C.H.U. D Angers, Angers
  - CH Louis Pasteur, Bagnols-sur-Cèze
  - Centre Medical Chateau Gaillard, Besançon
  - CH BESANCON - Hôpital Jean Minjoz, Besançon
  - Hopital Lapeyronie, Besançon
  - Polyclinique de Bois Bernard, Bois-Bernard
  - CHU Bordeaux, Bordeaux
  - CHU de Bordeaux - CHU Pellegrin, Bordeaux
  - Clinique Privé Jean Villar, Bruges
  - Clinique Saint Jean, Cagnes-sur-Mer
  - Clinique SAINT JEAN, Cagnes-sur-Mer
  - Hopital Prive Cannes Oxford, Cannes
  - Clinique Du Parc, Castelnau-le-Lez
  - Polyclinique Du Sidobre, Castres
  - Hopital Paul d'Egine, Champigny-sur-Marne
  - Hôpital Privé Paul d'Egine, Champigny-sur-Marne
  - Clinique des Cèdres, Cornebarrieu
  - Chu Henri Mondor, Créteil
  - Clinique Du Grand Large, Décines-Charpieu
  - CHRU Dijon le Bocage Central, Dijon
  - C.H.R.U. de Dijon, Dijon
  - Clinique de Fontiane Les Dijon, Dijon
  - Clinique Chirurgicale du Mail, La Rochelle
  - Clinique de Blanc Mesnil, Le Blanc-Mesnil
  - Hopital Bicetre (Ap-Hp), Le Kremlin-Bicêtre
  - Hopital Roger Salengro, Lille
  - Polyclinique Du Bois, Lille
  - Polyclinique Bordeaux Rive Droite, Lormont
  - Clinique Saint Charles, Lyon
  - Hopital P. Wertheimer, Lyon
  - Clinique Du Croise Laroche, Marcq-en-Barœul
  - APM La Timone, Marseille
  - Aphm Hopital de La Conception, Marseille
  - C.H.P. Clairval, Marseille
  - Hopital Européen, Marseille
  - Hôpital Privé Marsielle Beauregard, Marseille
  - CH Meulan - Les Mureaux, Meulan-en-Yvelines
  - Centre Aquitain du Dos, Mérignac
  - Hopital Lapeyronie, Montpellier
  - C.H.U. Nantes Hotel-Dieu, Nantes
  - Clinique Jules Verne, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - Cmc Ambroise Pare, Neuilly-sur-Seine
  - Clinique Saint-George, Nice
  - CHU de Nice - HOPITAL PASTEUR, Nice
  - CHU de Nice, Nice
  - Hôpital Privé les Franciscaines, Nîmes
  - G H U Caremeau, Nîmes
  - Hôpital les Franciscaines, Nîmes
  - Chr Orleans, Orléans
  - Groupe Hospitalier Paris St Joseph, Paris
  - Chu Pellegrin, Paris
  - Hopital Lariboisiere, Paris
  - Hopital Saint-Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Polyclinique Saint Martin, Pessac
  - Hopital Maison Blanche Chu Reims, Reims
  - Polyclinique Saint Andre, Reims
  - Hopital Charles Nicolle Chu Rouen, Rouen
  - Hôpital privé de la Loire, Saint-Etienne
  - Clinique Belledonne, Saint-Martin-d'Hères
  - Clinique Du Parc, Saint-Priest-en-Jarez
  - Nouvelle Clinique de l'Union, St.-Jean
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Polyclinique Du Parc, Toulouse
  - Clinique Medipole Garonne, Toulouse
  - Clinique de Vitrolles, Vitrolles